CLINICAL TRIAL: NCT01082965
Title: A Methodology Study To Evaluate The Acute Effects Of Donepezil On Regional Cerebral Perfusion And Cognition In Subjects With Amnestic MCI And Mild Alzheimer's Disease
Brief Title: Acute Effects Of Donepezil On Brain Perfusion And Memory In Subjects With Cognitive Impairment And Mild Alzheimer's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of slow enrollment. The decision to terminate the trial was not based on any safety or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: A9001437
Record Dates: First submitted 2010-02-26; First posted 2010-03-09 (Estimated); Results first posted 2013-09-12 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-07

CONDITIONS: Alzheimer's Disease
Keywords: ASL MRI; perfusion; cognition; donepezil; alzheimer's disease; translational medicine
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil — 5 mg tablets once daily for 7 days and then 10mg on 8th day
  Arms: Treatment
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
The study hypothesizes that donepezil will have a positive impact on brain blood flow deficits in subjects with memory deficits and/or mild dementia and that improvements in brain blood flow will be accompanied by improvements in memory.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and caregivers must provide written Informed Consent and be willing to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
* AD: Diagnostic evidence of probable AD consistent with Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) and National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria met by the site Physician at the time of the Screening visit. This evidence must be fully documented in the participant's file prior to the Baseline Visit.
* For amnestic Mild Cognitive Impairment (MCI): A Clinical Dementia Rating (CDR) of 0.5 (with memory box score of at least 0.5) and a memory complaint that is objectively verified using a test of episodic memory: Delayed recall from one paragraph of the Wechsler Logical Memory scale (cutoff scores by education - maximum score of 25).
* Less than or equal to 8 for 16 or more years of education; Less than or equal to 4 for 8-15 years of education; Less than or equal to 2 for 0-7 years of education.
* Mini Mental State Exam (MMSE) score of 21-30
* Male and female subjects of non child-bearing potential (or using appropriate birth control measures) who are at least 50 years of age.
* In generally good health, in the opinion of the Principal Investigator (PI), based on medical history, Body Mass Index (BMI), physical examination, vital signs, 12-lead ECG, and laboratory values, including hematology and chemistry values.
* No known genetic AD causes for early onset memory impairment (e.g., presenilin mutation), participants from a family with known autosomal dominant AD associated with mutations in APP, PS1, or PS2 genes or strongly suspected, but not yet identified mutations in APP, PS1 or PS2 genes or Down's syndrome are not eligible to enroll. Individuals from families with late onset AD with 2 or more affected family members may participate.

Type II diabetic subjects may be included provided that their disease and serum glucose values are controlled and being actively managed, as assessed by the PI using a fasting blood sugar and/or HgbA1C (per the PI's medical judgment in consultation with the Sponsor).

* Rosen-Modified Hachinski Ischemia Score less than or equal to 4.

Exclusion Criteria:

* Diagnosis or history of other possible cause for or significant contributor to dementia, including but not limited to other neurodegenerative disorders (eg, frontotemporal dementia, Lewy body disease, vascular dementia), vitamin B12 deficiency (reflex Methylmalonic Acid (MMA) and folate if B12 is low), untreated thyroid disease, syphilis, alcoholism, severe or recurrent head injury that is clinically relevant to the disease under study, or onset of dementia following heart surgery or cardiac arrest.
* Diagnosis or history of cerebrovascular disease (eg, stroke, transient ischemic attack), severe carotid stenosis, cerebral hemorrhage, intracranial tumor, subarachnoid hemorrhage, or subdural hematoma that could contribute to the subject's current cognitive or functional status, impair ability to fully participate in the trial or that may impact status during the one week study.
* Specific exclusionary brain MRI findings identified prior to study or at baseline as determined by the investigator that could either contribute to the subject's current cognitive or functional decline impair ability to fully participate in the trial or that may impact status during the trial:
* History of cancer within the last year (except for cutaneous basal cell, squamous cell cancer resolved by excision, colon polyp resolved by excision, or non-progressive prostate cancer per investigator's judgment).
* History of clinically significant cardiovascular or renal events.
* Subjects with uncontrolled hypertension even with therapeutic intervention
* History of clinically significant (as determined by the PI in consultation with the Sponsor) syncope, seizure, head trauma, or clinically significant unexplained loss of consciousness within the last 5 years.
* A diagnosis of major depressive disorder or other psychiatric illness as the primary diagnosis per the DSM-IV text revision (TR) criteria per the investigator's judgment.
* History of schizophrenia, bipolar disorder, or other severe mental illness.
* Known history of alcohol or drug abuse (as defined by the DSM-IV-TR) within 5 years prior to dosing or a positive result regarding use of illicit drugs on the drug screening test.
* History of clinically significant symptoms of pulmonary disease that requires treatment (eg. asthma, COPD, or other chronic respiratory conditions).
* Known positive Human immunodeficiency virus (HIV) status.
* Unwilling or unable to comply with the Life Style guidelines described in this protocol.

Exclusions Related to Medications or Procedures

* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) of Study Day 1.
* Use of tobacco- or nicotine-containing products within three months of study Day 1.

Use of medication(s) for cognitive enhancement ≤ 90 days before the first dose of study medication.

* Prescription: including but not limited to donepezil, galantamine, rivastigmine, tacrine, memantine, Axona™;
* Reason for stoppage of donepezil may not be related to tolerability issues or to gain entry in this study.
* Non-prescription treatments for cognitive enhancement.

  * Subjects with either non-removable ferromagnetic implants (such as cardiac pacemaker), aneurysm clips or other foreign bodies that would contraindicate a brain MRI scan.
  * A clinically significant (as determined by the PI) abnormality in the 12-lead ECG, including complete heart block, bradycardia (heart rate <40 beats/minute), sinus pauses >2 seconds, second or third degree heart block, QTc >450 or other abnormalities judged clinically significant by the PI.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001437&StudyName=Acute%20Effects%20Of%20Donepezil%20On%20Brain%20Perfusion%20And%20Memory%20In%20Subjects%20With%20Cognitive%20Impairment%20And%20Mild%20Alzheimer%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil: Donepezil 5 milligram (mg) tablet orally once daily up to Day 7, followed by donepezil 10 mg tablet orally once on Day 8.
- Placebo: Placebo matched to donepezil 5 mg tablet orally once daily up to Day 7, followed by placebo matched to donepezil 10 mg tablet orally once on Day 8.
Period: Overall Study
Arm/Group | Donepezil | Placebo
Started | 10 | 8
Completed | 9 | 6
Not Completed | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Donepezil: Donepezil 5 mg tablet orally once daily up to Day 7, followed by donepezil 10 mg tablet orally once on Day 8.
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 10 | 8 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 74.7 (9.6) | 70.6 (6.9) | 72.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Posterior Cingulate Cortex Perfusion at Hour 4 on Day 1
Description: Posterior cingulate cortex perfusion was measured by arterial spin labeling (ASL). ASL is a completely noninvasive magnetic resonance method to measure regional cerebral perfusion. Results are reported for average relative perfusion rate. Average relative perfusion rate is defined as the average absolute perfusion rate divided by the whole brain absolute perfusion rate at the same time point. Average absolute perfusion rate is the average of left absolute perfusion rate and right absolute perfusion rate at the same time point.
Time Frame: Baseline, 4 hours post-dose on Day 1
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of the study drug (donepezil or placebo). Here, 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 9 | 6
ratio
  Baseline | 1.243 (0.2586) | 1.564 (0.2494)
  Change at Hour 4 on Day 1 | 0.156 (0.5178) | -0.017 (0.3810)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Mixed model for repeated measures (MMRM) was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, Apolipoprotein E (ApoE) genotype, site as covariates; Test type: Superiority or Other; p = 0.9742, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; Leasts Square (LS) Mean = -0.01, 95% CI 2-sided [-0.60 to 0.58], Standard Error of Mean 0.265

2. Primary Outcome: Change From Baseline in Posterior Cingulate Cortex Perfusion at Hour 0 on Day 8
Description: Posterior cingulate cortex perfusion was measured by ASL. ASL is a completely noninvasive magnetic resonance method to measure regional cerebral perfusion. Results are reported for average relative perfusion rate. Average relative perfusion rate is defined as the average absolute perfusion rate divided by the whole brain absolute perfusion rate at the same time point. Average absolute perfusion rate is the average of left absolute perfusion rate and right absolute perfusion rate at the same time point.
Time Frame: Baseline, 1 minute post-dose (Hour 0) on Day 8
Population: FAS included all randomized participants who received at least 1 dose of the study drug (donepezil or placebo). Here, 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 9 | 6
ratio | 0.263 (0.4872) | 0.093 (0.5624)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.9638, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.01, 95% CI 2-sided [-0.51 to 0.49], Standard Error of Mean 0.232

3. Primary Outcome: Change From Baseline in Posterior Cingulate Cortex Perfusion at Hour 4 on Day 8
Description: as for outcome 2
Time Frame: Baseline, 4 hours post-dose on Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 9 | 6
ratio | -0.008 (0.2506) | -0.004 (0.3948)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2548, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.19, 95% CI 2-sided [-0.53 to 0.16], Standard Error of Mean 0.153

4. Secondary Outcome: Change From Baseline in Arterial Spin Label (ASL) Perfusion at Hour 4 on Day 1 and at Hour 0, 4 on Day 8
Description: Perfusion in anterior cingulate cortex, medial prefrontal cortex, precuneus, inferior parietal cortex and other regions of interest (whole brain gray, superior, medial and inferior temporal cortex; inferior and superior prefrontal cortex; insula, amygdala, thalamus, basal ganglia, hippocampus, Landau) was measured by ASL technique. ASL is a completely noninvasive magnetic resonance method to measure regional cerebral perfusion. Results are reported for relative perfusion rate. Relative perfusion rate is defined as the absolute perfusion rate divided by the whole brain absolute perfusion rate at the same time point.
Time Frame: Baseline, 4 hours post-dose on Day 1, 1 minute post-dose (Hour 0), 4 hours post-dose on Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 9 | 6
ratio
  Baseline: Whole Brain Gray | 1.486 (0.1215) | 1.500 (0.0869)
  Baseline: Superior Temporal Cortex | 1.749 (0.2774) | 1.773 (0.1732)
  Baseline: Medial Temporal Cortex | 1.753 (0.3186) | 1.718 (0.2778)
  Baseline: Inferior Temporal Cortex | 1.260 (0.4634) | 1.173 (0.4024)
  Baseline: Medial Prefrontal Cortex | 1.488 (0.1830) | 1.709 (0.1441)
  Baseline: Inferior Prefrontal Cortex | 1.381 (0.2205) | 1.486 (0.1673)
  Baseline: Superior Prefrontal Cortex | 1.308 (0.1236) | 1.443 (0.2046)
  Baseline: Inferior Parietal Cortex | 1.610 (0.2824) | 1.714 (0.1628)
  Baseline: Insula | 1.390 (0.1785) | 1.533 (0.2130)
  Baseline: Precuneus | 1.357 (0.1904) | 1.505 (0.2781)
  Baseline: Anterior Cingulate Cortex | 1.236 (0.2265) | 1.442 (0.1753)
  Baseline: Amygdala | 1.067 (0.3025) | 1.256 (0.2966)
  Baseline: Thalamus | 1.417 (0.4886) | 1.468 (0.3061)
  Baseline: Basal Ganglia | 1.120 (0.2781) | 1.241 (0.2461)
  Baseline: Hippocampus | 1.327 (0.2726) | 1.389 (0.1229)
  Baseline: Landau | 1.916 (0.3753) | 2.025 (0.0940)
  Change at Hour 4 on Day 1: Whole Brain Gray | 0.018 (0.2309) | 0.050 (0.1010)
  Change at Hour 4 on Day 1:Superior Temporal Cortex | 0.031 (0.3430) | 0.023 (0.3002)
  Change at Hour 4 on Day 1: Medial Temporal Cortex | -0.066 (0.5297) | -0.006 (0.2549)
  Change at Hour 4 on Day 1:Inferior Temporal Cortex | -0.052 (0.6289) | 0.090 (0.2734)
  Change at Hour 4 on Day 1:Medial Prefrontal Cortex | 0.035 (0.2704) | -0.164 (0.2054)
  Change at Hour4 on Day1:Inferior Prefrontal Cortex | 0.143 (0.1987) | -0.061 (0.2299)
  Change at Hour4 on Day1:Superior Prefrontal Cortex | 0.064 (0.2702) | -0.062 (0.2361)
  Change at Hour 4 on Day 1:Inferior Parietal Cortex | -0.054 (0.2411) | -0.016 (0.1848)
  Change at Hour 4 on Day 1: Insula | 0.154 (0.2813) | 0.096 (0.3276)
  Change at Hour 4 on Day 1: Precuneus | -0.024 (0.3002) | 0.053 (0.2952)
  Change at Hour 4 on Day1:Anterior Cingulate Cortex | 0.118 (0.2168) | 0.173 (0.2709)
  Change at Hour 4 on Day 1: Amygdala | 0.187 (0.5504) | 0.175 (0.3785)
  Change at Hour 4 on Day 1: Thalamus | 0.244 (0.5697) | -0.038 (0.2209)
  Change at Hour 4 on Day 1: Basal Ganglia | 0.292 (0.4557) | 0.014 (0.1761)
  Change at Hour 4 on Day 1: Hippocampus | 0.128 (0.2115) | 0.036 (0.2915)
  Change at Hour 4 on Day 1: Landau | -0.051 (0.3923) | -0.033 (0.1952)
  Change at Hour 0 on Day 8: Whole Brain Gray | 0.058 (0.1024) | 0.028 (0.1569)
  Change at Hour 0 on Day 8:Superior Temporal Cortex | 0.051 (0.2678) | 0.038 (0.3095)
  Change at Hour 0 on Day 8: Medial Temporal Cortex | -0.015 (0.3095) | -0.052 (0.2575)
  Change at Hour 0 on Day 8:Inferior Temporal Cortex | 0.084 (0.6856) | -0.012 (0.3842)
  Change at Hour 0 on Day 8:Medial Prefrontal Cortex | -0.198 (0.4168) | -0.173 (0.3050)
  Change at Hour0 on Day8:Inferior Prefrontal Cortex | 0.043 (0.3353) | 0.010 (0.2188)
  Change at Hour0 on Day8:Superior Prefrontal Cortex | -0.152 (0.3120) | -0.019 (0.2863)
  Change at Hour 0 on Day 8:Inferior Parietal Cortex | 0.005 (0.5185) | -0.106 (0.2009)
  Change at Hour 0 on Day 8: Insula | 0.103 (0.2679) | 0.154 (0.1816)
  Change at Hour 0 on Day 8: Precuneus | 0.055 (0.4065) | 0.059 (0.3475)
  Change at Hour 0 on Day8:Anterior Cingulate Cortex | 0.279 (0.4424) | 0.167 (0.3681)
  Change at Hour 0 on Day 8: Amygdala | 0.170 (0.5388) | 0.083 (0.4233)
  Change at Hour 0 on Day 8: Thalamus | 0.195 (0.6486) | -0.063 (0.4992)
  Change at Hour 0 on Day 8: Basal Ganglia | 0.243 (0.3925) | 0.040 (0.3106)
  Change at Hour 0 on Day 8: Hippocampus | 0.170 (0.2832) | 0.047 (0.2551)
  Change at Hour 0 on Day 8: Landau | -0.030 (0.5354) | -0.105 (0.2642)
  Change at Hour 4 on Day 8: Whole Brain Gray | 0.010 (0.1286) | -0.022 (0.0945)
  Change at Hour 4 on Day 8:Superior Temporal Cortex | 0.126 (0.3065) | -0.037 (0.1319)
  Change at Hour 4 on Day 8: Medial Temporal Cortex | -0.103 (0.2852) | -0.110 (0.2551)
  Change at Hour 4 on Day 8:Inferior Temporal Cortex | -0.194 (0.5644) | -0.102 (0.3114)
  Change at Hour 4 on Day 8:Medial Prefrontal Cortex | 0.111 (0.3606) | -0.038 (0.2262)
  Change at Hour4 on Day8:Inferior Prefrontal Cortex | -0.031 (0.2477) | -0.001 (0.2342)
  Change at Hour4 on Day8:Superior Prefrontal Cortex | 0.225 (0.3460) | -0.007 (0.1348)
  Change at Hour 4 on Day 8:Inferior Parietal Cortex | -0.175 (0.4557) | -0.017 (0.1560)
  Change at Hour 4 on Day 8: Insula | 0.148 (0.1477) | 0.078 (0.2317)
  Change at Hour 4 on Day 8: Precuneus | -0.110 (0.3846) | 0.074 (0.3035)
  Change at Hour 4 on Day8:Anterior Cingulate Cortex | 0.180 (0.2939) | 0.062 (0.1423)
  Change at Hour 4 on Day 8: Amygdala | 0.097 (0.4984) | 0.019 (0.3100)
  Change at Hour 4 on Day 8: Thalamus | -0.124 (0.5028) | -0.077 (0.5330)
  Change at Hour 4 on Day 8: Basal Ganglia | 0.084 (0.3393) | -0.066 (0.2787)
  Change at Hour 4 on Day 8: Hippocampus | 0.041 (0.2770) | 0.017 (0.1225)
  Change at Hour 4 on Day 8: Landau | -0.208 (0.3152) | 0.008 (0.1418)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Whole Brain Gray: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6316, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.03, 95% CI 2-sided [-0.18 to 0.12], Standard Error of Mean 0.057
Statistical Analysis 2: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Whole Brain Gray: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6256, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.03, 95% CI 2-sided [-0.12 to 0.19], Standard Error of Mean 0.063
Statistical Analysis 3: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Whole Brain Gray: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.5847, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.03, 95% CI 2-sided [-0.12 to 0.19], Standard Error of Mean 0.059
Statistical Analysis 4: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Superior Temporal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.1555, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.19, 95% CI 2-sided [-0.46 to 0.09], Standard Error of Mean 0.123
Statistical Analysis 5: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Superior Temporal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.2416, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.18, 95% CI 2-sided [-0.51 to 0.14], Standard Error of Mean 0.151
Statistical Analysis 6: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Superior Temporal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.8070, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.03, 95% CI 2-sided [-0.33 to 0.26], Standard Error of Mean 0.134
Statistical Analysis 7: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Medial Temporal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6828, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.08, 95% CI 2-sided [-0.59 to 0.43], Standard Error of Mean 0.189
Statistical Analysis 8: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Medial Temporal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.8987, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.01, 95% CI 2-sided [-0.26 to 0.29], Standard Error of Mean 0.109
Statistical Analysis 9: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Medial Temporal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.8922, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.02, 95% CI 2-sided [-0.28 to 0.25], Standard Error of Mean 0.117
Statistical Analysis 10: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Inferior Temporal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.7555, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.07, 95% CI 2-sided [-0.39 to 0.52], Standard Error of Mean 0.203
Statistical Analysis 11: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Inferior Temporal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.1928, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.30, 95% CI 2-sided [-0.18 to 0.79], Standard Error of Mean 0.218
Statistical Analysis 12: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Inferior Temporal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.4946, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.12, 95% CI 2-sided [-0.26 to 0.49], Standard Error of Mean 0.161
Statistical Analysis 13: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Medial Prefrontal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.7029, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.08, 95% CI 2-sided [-0.56 to 0.40], Standard Error of Mean 0.196
Statistical Analysis 14: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Medial Prefrontal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.1085, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.30, 95% CI 2-sided [-0.68 to 0.08], Standard Error of Mean 0.171
Statistical Analysis 15: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Medial Prefrontal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.3588, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.13, 95% CI 2-sided [-0.44 to 0.18], Standard Error of Mean 0.132
Statistical Analysis 16: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Inferior Prefrontal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.3053, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.17, 95% CI 2-sided [-0.20 to 0.53], Standard Error of Mean 0.151
Statistical Analysis 17: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Inferior Prefrontal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.9861, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.00, 95% CI 2-sided [-0.36 to 0.36], Standard Error of Mean 0.160
Statistical Analysis 18: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Inferior Prefrontal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6558, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.07, 95% CI 2-sided [-0.41 to 0.28], Standard Error of Mean 0.140
Statistical Analysis 19: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Superior Prefrontal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.9471, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.01, 95% CI 2-sided [-0.53 to 0.51], Standard Error of Mean 0.145
Statistical Analysis 20: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Superior Prefrontal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.2136, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.27, 95% CI 2-sided [-0.77 to 0.23], Standard Error of Mean 0.186
Statistical Analysis 21: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Superior Prefrontal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6435, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.10, 95% CI 2-sided [-0.47 to 0.67], Standard Error of Mean 0.189
Statistical Analysis 22: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Inferior Parietal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.0659, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.20, 95% CI 2-sided [-0.41 to 0.02], Standard Error of Mean 0.086
Statistical Analysis 23: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Inferior Parietal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.7687, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.05, 95% CI 2-sided [-0.41 to 0.31], Standard Error of Mean 0.158
Statistical Analysis 24: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Inferior Parietal Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.1061, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.32, 95% CI 2-sided [-0.73 to 0.10], Standard Error of Mean 0.163
Statistical Analysis 25: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Insula: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.3925, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.11, 95% CI 2-sided [-0.41 to 0.19], Standard Error of Mean 0.124
Statistical Analysis 26: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Insula: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.1991, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.22, 95% CI 2-sided [-0.58 to 0.14], Standard Error of Mean 0.161
Statistical Analysis 27: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Insula: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.5176, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.10, 95% CI 2-sided [-0.45 to 0.24], Standard Error of Mean 0.151
Statistical Analysis 28: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Precuneus: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.3140, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.16, 95% CI 2-sided [-0.50 to 0.18], Standard Error of Mean 0.143
Statistical Analysis 29: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Precuneus: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6348, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.08, 95% CI 2-sided [-0.46 to 0.29], Standard Error of Mean 0.171
Statistical Analysis 30: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Precuneus: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.1491, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.26, 95% CI 2-sided [-0.64 to 0.12], Standard Error of Mean 0.165
Statistical Analysis 31: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Anterior Cingulate Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.4226, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.16, 95% CI 2-sided [-0.59 to 0.27], Standard Error of Mean 0.192
Statistical Analysis 32: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Anterior Cingulate Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.9778, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.01, 95% CI 2-sided [-0.49 to 0.50], Standard Error of Mean 0.228
Statistical Analysis 33: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Anterior Cingulate Cortex: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.9456, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.01, 95% CI 2-sided [-0.40 to 0.43], Standard Error of Mean 0.179
Statistical Analysis 34: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Amygdala: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.2299, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.20, 95% CI 2-sided [-0.55 to 0.15], Standard Error of Mean 0.162
Statistical Analysis 35: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Amygdala: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.5069, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.13, 95% CI 2-sided [-0.54 to 0.28], Standard Error of Mean 0.188
Statistical Analysis 36: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Amygdala: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.3524, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.14, 95% CI 2-sided [-0.45 to 0.17], Standard Error of Mean 0.143
Statistical Analysis 37: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Thalamus: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.4182, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.34, 95% CI 2-sided [-0.80 to 1.47], Standard Error of Mean 0.358
Statistical Analysis 38: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Thalamus: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.3630, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.31, 95% CI 2-sided [-0.42 to 1.04], Standard Deviation 0.326
Statistical Analysis 39: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Thalamus: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.9837, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.01, 95% CI 2-sided [-0.73 to 0.74], Standard Error of Mean 0.263
Statistical Analysis 40: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Basal Ganglia: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.0974, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.19, 95% CI 2-sided [-0.04 to 0.42], Standard Error of Mean 0.102
Statistical Analysis 41: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Basal Ganglia: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.1246, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.11, 95% CI 2-sided [-0.04 to 0.27], Standard Error of Mean 0.067
Statistical Analysis 42: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Basal Ganglia: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6190, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.06, 95% CI 2-sided [-0.20 to 0.32], Standard Error of Mean 0.119
Statistical Analysis 43: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Hippocampus: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6350, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.07, 95% CI 2-sided [-0.39 to 0.25], Standard Error of Mean 0.140
Statistical Analysis 44: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Hippocampus: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.8205, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.04, 95% CI 2-sided [-0.40 to 0.32], Standard Error of Mean 0.164
Statistical Analysis 45: Comparison: Donepezil; Change at Hour 4 on Day 8, Hippocampus: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.2959, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.15, 95% CI 2-sided [-0.42 to 0.14], Standard Error of Mean 0.123
Statistical Analysis 46: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 1, Landau: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.5520, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.12, 95% CI 2-sided [-0.56 to 0.32], Standard Error of Mean 0.194
Statistical Analysis 47: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Landau: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.9046, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.03, 95% CI 2-sided [-0.50 to 0.45], Standard Error of Mean 0.220
Statistical Analysis 48: Comparison: Donepezil vs Placebo; Change at Hour 4 on Day 8, Landau: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.0402, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -0.32, 95% CI 2-sided [-0.62 to -0.02], Standard Error of Mean 0.125

5. Secondary Outcome: Change From Baseline in CogState Continuous Paired Associate Learning (CPAL) at Hour 5 on Day 1 and at Hour 1, 5 on Day 8
Description: CPAL: a cognitive test which assessed visual episodic learning. Participant was to learn and remember picture locations on the screen and was to tap the target on the central location to begin. As each picture was revealed, the participant was to remember where the picture was located and tap that location. After 4 pictures were placed correctly, second round started. In second round pictures remain in the same locations, but their order of presentation in the center of the screen was different to that of the first round (randomized). The same process was repeated for round 3 and round 4. The outcome was the number of errors made in correctly placing each of the 4 patterns in their location 4 times.
Time Frame: Baseline, 5 hours post-dose on Day 1; 1, 5 hours post-dose on Day 8
Population: FAS included all randomized participants who received at least 1 dose of the study drug (donepezil or placebo). Here, 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure. n=participants who were evaluable at specified time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 9 | 8
errors
  Baseline (n=9, 8) | 46.222 (28.7436) | 37.625 (17.8641)
  Change at Hour 5 on Day 1 (n=9, 8) | 4.333 (24.0936) | -2.625 (28.9084)
  Change at Hour 1 on Day 8 (n=9, 6) | -5.444 (31.9653) | -15.833 (15.8293)
  Change at Hour 5 on Day 8 (n=9, 6) | 2.000 (16.3325) | -8.000 (17.4126)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Change at Hour 5 on Day 1: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6880, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 5.00, 95% CI 2-sided [-21.82 to 31.82], Standard Error of Mean 12.110
Statistical Analysis 2: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.3157, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 9.79, 95% CI 2-sided [-11.30 to 30.87], Standard Error of Mean 9.143
Statistical Analysis 3: Comparison: Donepezil vs Placebo; Change at Hour 5 on Day 8: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.3228, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 9.86, 95% CI 2-sided [-13.56 to 33.28], Standard Error of Mean 8.921

6. Secondary Outcome: Change From Baseline in Rey Auditory Verbal Learning Test (RAVLT): Immediate and Delayed Recall at Hour 5 on Day 8
Description: RAVLT, in immediate recall (IR) list of 15 words (list A) was read aloud to participant 5 times followed by a test of spontaneous retrieval (A1 to A5). After fifth attempt a list of interference, comprising 15 words (list B) was read to participant followed by its retrieval (B1). After attempt B1 examiner asked individual to recall words from list A, without reading it again (A6). Score range: 0-105, higher scores=less impairment. Delayed recall (DR):after a 20-minute interval examiner asked individual to remember words from list A without reading this list; in recognition performance a list comprising 15 words from list A, 15 words from list B, 20 distracting words (similar to words in list A, B) was read to individual. Upon each word read aloud, individual asked to indicate if it belonged to list A, or not. Score range: 0-30, higher scores=less impairment.
Time Frame: Baseline, 5 hours post-dose on Day 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale
  Baseline: Total IR (n=9, 8) | 25.667 (7.3144) | 27.000 (9.3960)
  Baseline: Total DR (n=9, 8) | 2.444 (2.3511) | 2.375 (2.1998)
  Change at Hour 5 on Day 8:Total IR (n=9, 6) | 3.333 (4.1833) | 5.667 (4.3665)
  Change at Hour 5 on Day 8: Total DR (n=9, 6) | 0.444 (1.9437) | 0.333 (3.0111)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Total IR: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.2540, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = -4.39, 95% CI 2-sided [-12.90 to 4.12], Standard Error of Mean 3.479
Statistical Analysis 2: Comparison: Donepezil vs Placebo; Total DR: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.7684, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.60, 95% CI 2-sided [-4.17 to 5.37], Standard Error of Mean 1.950

7. Secondary Outcome: Change From Baseline in CogState Test Battery at Hour 5 on Day 1 and at Hour 0, 5 on Day 8
Description: Computerized test battery used to assess detection and identification task. CogState detection task: a measure of simple reaction time, provided valid assessment of psychomotor function. Participants were required to press a "YES" response key as soon as they detected an event (a card turning face up presented in center of the computer screen). The software measured the response time to detect each event. CogState identification task: measure of choice reaction time, provided a valid assessment of visual attention. Participants were required to decide "YES" or "NO" as to whether the event met a predefined and unchanging criterion (is the color of the card red?) while the event (a card turning face up) occurred in the center of the computer screen. The software measured the speed and accuracy of each response.
Time Frame: Baseline, 5 hours post-dose on Day 1; 1, 5 hours post-dose on Day 8
Population: FAS included all randomized participants who received at least 1 dose of the study drug (donepezil or placebo). Here, 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure. n=participants who were evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: log10 milliseconds
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 9 | 8
log10 milliseconds
  Baseline: Detection Task (n=9, 8) | 2.572 (0.1192) | 2.542 (0.0953)
  Baseline: Identification Task (n=9, 8) | 2.708 (0.0635) | 2.727 (0.0540)
  Change at Hour 5 on Day 1: Detection Task (n=9, 8) | 0.002 (0.0931) | 0.024 (0.0706)
  Change at Hour5 on Day1:Identification Task(n=9,8) | 0.020 (0.0355) | 0.012 (0.0371)
  Change at Hour 0 on Day 8: Detection Task (n=9, 6) | 0.004 (0.1184) | -0.032 (0.0512)
  Change at Hour0 on Day8:Identification Task(n=9,6) | 0.005 (0.0630) | 0.004 (0.0493)
  Change at Hour 5 on Day 8: Detection Task (n=9, 6) | -0.005 (0.1001) | 0.004 (0.0508)
  Change at Hour5 on Day8:Identification Task(n=9,6) | 0.034 (0.0782) | 0.004 (0.0625)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Change at Hour 5 on Day 1, Detection Task: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.4940, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.04, 95% CI 2-sided [-0.09 to 0.17], Standard Error of Mean 0.059
Statistical Analysis 2: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Detection Task: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.1031, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.10, 95% CI 2-sided [-0.02 to 0.22], Standard Error of Mean 0.057
Statistical Analysis 3: Comparison: Donepezil vs Placebo; Change at Hour 5 on Day 8, Detection Task: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.3277, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.05, 95% CI 2-sided [-0.06 to 0.16], Standard Error of Mean 0.048
Statistical Analysis 4: Comparison: Donepezil; Change at Hour 5 on Day 1, Identification Task: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.6585, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.01, 95% CI 2-sided [-0.05 to 0.08], Standard Error of Mean 0.029
Statistical Analysis 5: Comparison: Donepezil vs Placebo; Change at Hour 0 on Day 8, Identification Task: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.8863, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.00, 95% CI 2-sided [-0.07 to 0.08], Standard Error of Mean 0.033
Statistical Analysis 6: Comparison: Donepezil vs Placebo; Change at Hour 5 on Day 8, Identification Task: MMRM was used with treatment, time, treatment-by-time interaction as fixed effects and baseline, age, gender, ApoE genotype, site as covariates; Test type: Superiority or Other; p = 0.4388, Mixed Models Analysis — Statistical significance level alpha (2-sided) was 0.05; LS Mean Difference = 0.04, 95% CI 2-sided [-0.06 to 0.13], Standard Error of Mean 0.044

ADVERSE EVENTS:
Arm/Group | Donepezil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 3/10 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil (N=10) | Placebo (N=8)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated because of the prohibitively low recruitment rate and the reassessment of the Neuroscience Research Unit portfolio. The decision to terminate the study was not based on any safety or efficacy concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.